## Study Protocol and Statistical Analysis Plan (SAP)

# The Effects of Weight Science and Nutrition Education on Weight Control Beliefs, Body Image, Self-Esteem and Eating Patterns in Undergraduate Dieters

Unique Protocol ID #19334

November 4th, 2025

**Authors:** Keisha Gobin, Ph.D., C.Psych<sup>1</sup>

Sarah Potter, B.A., Graduate Student<sup>2</sup>

Mindy Tat, B.Sc. (Hons) (Expected 2026)<sup>3</sup>

**Program:** 1. Assistant Professor, Department of Psychiatry and Behavioral

Neurosciences, McMaster University, Hamilton, Canada and Co-Clinical Lead, Eating Disorders Clinic, St Joseph's Healthcare,

Hamilton, Canada

2. Graduate student, Department of Psychology, Neuroscience, and Behavior, McMaster University, Hamilton, Ontario, Canada and Eating Disorders Clinic, St. Joseph's Healthcare Hamilton, Hamilton,

Ontario, Canada

3. Thesis student, Department of Psychology, Neuroscience and

Behavior, McMaster University, Hamilton, Canada

#### **Abstract**

# Background

Individuals who engage in dieting behaviours are at elevated risk for developing disordered eating and eating disorders (Stice et al., 2017; Barakat et al., 2023; Jebeile et al., 2019). These individuals have a belief that weight is within their control and, as such, are likely to engage in unhealthy weight control practices associated with poor psychological well-being (Neumark-Sztainer et al., 2007; Kabakuş & Bilici, 2022). Research suggests two weight control beliefs: (1) the belief in controlling one's weight and (2) the belief in controlling one's lifestyle with acceptance of the resulting weight (Laliberte et al., 2007). In non-clinical samples, the belief in controlling one's weight is positively associated with disordered eating, body dissatisfaction and poor self-esteem (Laliberte et al., 2007). Meanwhile, the belief in controlling one's lifestyle with acceptance of the resulting weight is *negatively* associated with disordered eating, body dissatisfaction and poor self-esteem (Laliberte et al., 2007). Providing weight science education to non-dieters has been shown to significantly decrease the belief in controlling one's weight and increase the belief in controlling one's lifestyle with acceptance of the resulting weight (Laliberte et al., 2014). However, the effect size for the belief in controlling one's lifestyle with acceptance of the resulting weight was small (Laliberte et al., 2014). Given the risks to those who diet, it is essential to investigate whether providing education about weight science and healthy lifestyle practices specifically benefits this group.

#### Objectives:

This study investigates whether providing information on healthy eating and weight science will result in a significant and meaningful change to both belief in controlling one's weight and belief in controlling one's lifestyle with acceptance of the resulting weight. The study also investigates whether a change in weight control beliefs will predict a change in one's intent to diet, self-esteem, dietary restraint, and body appreciation. Given that individuals who endorse dieting behaviours are at a substantially greater risk for developing disordered eating and eating disorders, the present study will exclusively recruit individuals who self-identify as currently dieting, to explore whether providing this education may be beneficial for this specific high-risk group.

#### **Implications**

This study will evaluate the effects of two educational components designed to influence weight control beliefs and related risk factors for eating disorders, including dietary restraint, the intent to diet, body dissatisfaction, and self-esteem, among individuals who diet. By examining how psychoeducation impacts these outcomes, the study aims to provide insights that could inform future interventions for populations at higher risk of developing eating disorders. Additionally, the findings may shed light on the potential benefits of specific psychoeducational components commonly used in cognitive-behavioural therapy for eating disorder populations.

#### Study purpose and rationale

Background:

In North America, body dissatisfaction and fear of being "fat" are common experiences reported by women (Ackard et al., 2007; Cash et al., 2004; Piran & Gadalla, 2007). A review conducted in 2004 found that 29% of white college-age women report extreme body dissatisfaction, and a different large-scale study found 26% of Canadian women report a strong fear of being fat (Cash et al., 2004; Piran & Gadalla, 2007). These findings are concerning given that body dissatisfaction is a risk factor for the development and maintenance of disordered eating (Polivy & Herman, 2002; Stice & Shaw, 2002). As a result of body dissatisfaction, women often engage in dieting behaviours to try and change the shape of their body. A study on college women found that 82% of women in college use at least one dieting behaviour daily, and 33% of them also engage in more extreme strategies to control their weight, like using laxatives or vomiting, monthly (Mintz & Betz, 1988). Recent research further asserts that dieting predicts the onset of eating disorder symptoms across multiple populations and follow-up periods (Stice et al., 2017; Patton et al., 1990; Jebeile et al., 2019), and that dieting behaviours among university students remain prevalent and are associated with unhealthy eating patterns and eating disorder risk (Kabakus & Bilici, 2022). Furthermore, individuals who diet may hold stronger beliefs in controlling their weight (Vartanian & Herman, 2006), potentially placing them at greater risk for disordered eating outcomes. By focusing exclusively on dieters in this study, we can explore whether education about weight science can alter maladaptive beliefs.

One such set of maladaptive beliefs that may place dieters at increased risk involves their beliefs about weight control itself. Specifically, research suggests that individuals tend to hold one of two primary beliefs about weight control: (1) the belief in personal control over one's weight and (2) the belief in controlling one's lifestyle with acceptance of the resulting weight (Laliberte et al., 2007). In non-clinical samples, the belief in controlling one's weight is positively associated with disordered eating, body dissatisfaction and poor self-esteem (Laliberte et al., 2007). In contrast, the belief in controlling one's lifestyle with acceptance of the resulting weight is *negatively* associated with disordered eating, body dissatisfaction and poor self-esteem (Laliberte et al., 2007). Providing weight science education has been shown to significantly (with large effect size) decrease the belief in personal control over one's weight. Weight science education also significantly increased the belief in controlling one's lifestyle with acceptance of the resulting weight (Laliberte et al., 2014); however, the effect size for the belief in controlling one's lifestyle with acceptance of the resulting weight was small (Laliberte et al., 2014). Of interest, only the small increase in the belief in controlling one's lifestyle with weight acceptance predicted positive changes in body dissatisfaction, self-esteem and measures of disordered eating.

In cognitive behaviour therapy (CBT) for eating disorders, it is common for weight science teaching to be supported by information on healthy eating (Fairburn, 2008); and there is research in clinical settings demonstrating that CBT results in a decrease in the belief in personal control over weight, and an increase in the belief in striving for a healthy lifestyle with weight

acceptance (Laliberte & Lucibello, 2022). In the present study, we propose to extend the previous study on the effects of education on weight control beliefs in a non-clinical setting by examining the effects of weight control and nutrition education among undergraduate gender-based women who are dieting. Our objective is to determine whether the two components together are more effective in changing weight control beliefs than either alone.

#### *Hypothesis:*

# We expect:

- 1. Weight science education alone will decrease belief in personal control over weight but will have little to no effect on belief in choosing a healthy lifestyle/weight acceptance.
- 2. Nutrition education alone will increase belief in choosing a healthy lifestyle/weight acceptance but will have little to no effect on the belief in personal control over weight.
- 3. Weight science and nutrition teaching combined will both decrease the belief of personal control over weight and an increase the belief in choosing a healthy lifestyle/weight acceptance.
- 4. Change in weight control beliefs will predict changes in body appreciation, the intent to diet, self-esteem, and dietary restraint.

# Description of the population to be studied, inclusion and exclusion criteria

As disordered eating and negative body image are prevalent in gender-based women in early adulthood, a sample of non-clinical undergraduate students, who self-identify as women, will be recruited to participate in the study. Additionally, given that dieting is a well-established risk factor for the development of eating disorders, only participants who self-identify as currently engaging in dieting behaviours—for the purposes of weight loss—will be eligible for participation. Participants with who do not have normal hearing (or corrected to normal hearing) or vision (or corrected to normal vision) will not be eligible for this study due to the audio-visual nature of the interventions and questionnaires. All participants will be recruited via the SONA platform, an online recruitment site for students and faculty in the PNB Department at McMaster University. The SONA pre-screen self-report questionnaire will be used to assess eligibility for this criteria.

#### *Inclusion Criteria*:

A participant will be eligible to participate in the study if they meet the following criteria based on the SONA pre-screen questionnaire:

- 1. 18 years of age or older
- 2. A female or trans-female gender identity
- 3. Be restricting their eating to try and lose weight

- 4. Normal or correct-to-normal visual acuity
- 5. Normal or correct-to-normal auditory acuity

The SONA pre-screen self-report questionnaire is set-up and managed by the PNB Department. It is completed by all potential participants when they sign up for a SONA account. It is used to filter research studies such that participants can only view advertisements for studies they are eligible to participate in. Eligibility is determined solely through the SONA pre-screen system. Study investigators do not design or influence the pre-screen questions, response options, or eligibility logic, and do not have access to any data collected in the pre-screening process. No pre-screen information will be retained or used as part of this study. At the sign-up stage, participants are able to select a date/time to complete the study at their convenience.

It should be noted that SONA has a limited number of items that researchers can use for the purpose of pre-screening potential study participants. Given that some individuals may accidentally bypass the eligibility criteria on the SONA pre-screen questionnaire, we included a Screener instrument on our REDCap survey to ensure that participants are restricting their eating to try and lose weight. If participants do not endorse dieting, they will be redirected to the end of the study; however, they will still receive credit for participating.

#### Sample size (and how sample size was determined)

The sample size was determined using a power analysis for ANOVA conducted in R Studio. An effect size of 0.25 was used to conduct the power analysis. The effect size is a conservative estimate based on the results of a similar study conducted by Laliberte et al. 2014. The results of the power analysis recommend 53 participants in each study condition, resulting in a total of 159 participants overall.

```
pwr.anova.test(k=3, n=NULL, f=0.25, sig.level = 0.05, power=0.8) 
Output: Balanced one-way analysis of variance power calculation k = 3
n = 52.3966
f = 0.25
sig.level = 0.05
power = 0.8
NOTE: n is number in each group
```

There is a maximum of 15 participants per group, as the rooms available can accommodate up to 15 people. To ensure an equal number of participants in each condition, we will conduct 10-12 groups, each comprising of 10-15 participants. This will result in approximately 50 participants in each condition, and a total of 150 participants in the experiment. The experimental conditions will be randomly assigned to groups, ensuring equal representation of experimental conditions

across academic semesters. An additional consideration when determining the sample size was the limitation imposed by the Department of Psychology, Neuroscience and Behaviour. The department restricts researchers to a maximum of 150 credits per term. Since participants earn one credit for every hour of participation, this two-hour experiment grants them two credits. Due to this policy, a maximum of 75 students can be enrolled in the study per term, allowing data to be collected from a total of 150 students over two academic semesters.

#### Design and detailed description of methodology

Design:

Each group of participants will be randomly assigned to one of three conditions: 1) weight science + control (sleep education); 2) control (sleep education) + healthy eating education; or 3) weight science + healthy eating education. The sleep education module serves as a neutral placebo control condition, designed to provide participants with general, non-weight-related educational content. It is not expected to influence any of the study's primary outcomes related to dieting intentions, eating behaviours, body image, or self-esteem.

Participants will have the opportunity to self-select from the available timeslots for the study, with each timeslot accommodating a maximum of 15 participants, resulting in approximately 10 clusters for a total sample size of 150. Subsequently, each group of students will be randomly assigned to one of the experimental conditions. Prior to data collection, a lab mate who is not involved in participant recruitment, data collection, or analysis will generate the randomization sequence (e.g., alternating Condition 1, Condition 2, and Condition 3 in a random order) using a random number generator. Each session will then be pre-assigned to one of the three intervention conditions based on this randomization schedule. The lead investigator will be informed of the assigned condition only on the day of the session to ensure that participant assignment remains fully random and that blinding is maintained in advance, minimizing any potential anticipatory or selection bias.

The study is scheduled to be conducted from January 2026 to August 2026. This timeline aligns with the policy set forth by the Department of Psychology, Neuroscience, and Behavior, which restricts researchers to a maximum of 150 credits per term.

# Procedure:

After a participant completes the study sign-up procedure, they will select a time and date to complete the study in person at McMaster University in the Psychology Building. We have requested in the advertisement that participants bring a device (i.e., cellphone, laptop, tablet) to complete the online consent form and questionnaires. A reminder email will be sent 24 hours before the participants' scheduled study session, reminding them to bring a device. If any participant does not have access to a device, we will provide a spare tablet for the participant to access the consent form and study questionnaires.

Once participants have signed up for the study via SONA, they will receive the room number and detailed directions on how to reach the designated location. The student investigator

will be present at the pre-specified time and location to meet the participant. Furthermore, 24 hours prior to the study session, participants will receive a reminder email. This email will include the date, time and location of the study location, as well as a reminder to participants to bring, if possible, an electronic device such as their phone, laptop or tablet.

Once the participant arrives at the in-person study location, they will receive access to a link via SONA to sign an online consent form via REDCap. The participant can ask any questions about the study prior to signing the consent form to the student investigator in the room. If the participant agrees to participate in the study, they will be required to provide their full name, electronic signature, and the date to indicate their informed consent. Participants will be required to check a box indicating that they have had the opportunity to ask any questions that they may have about the study to ensure that participants are aware of and have accessed (as needed) the research team to clarify any questions. If a participant provides their informed consent, they will be directed to a page where they are able to download a copy of their signed consent form.

Once consent is obtained, the participants will answer some preliminary questions. All study questionnaires will be completed using REDCap. The first two questions in the experiment ask the participant to input their McMaster email and student number. These questions are required before the participant can continue with the experiment. The information will be used to provide them with course credit for the study. Additionally, the email provided will be used by the research team to ensure that all participants receive a copy of the consent form that includes both the participant's and investigator's signatures. Once a participant has signed the consent form, the lead Student Investigator (Mindy Tat) will download a copy of the signed consent form into the secure internal network of McMaster University. At this stage, the lead Student Investigator will provide her electronic signature on the consent form using Adobe Reader (on the McMaster internal network). The completed consent form will then be emailed to the participant via encrypted email, offered through McMaster Outlook. This will occur within 24 hours of the participant providing their consent.

After completing the screener and consent form, participants will be automatically redirected to the study questionnaires. Participants will begin by completing the following questionnaires in REDCap: demographic questionnaire, Three-Factor Eating Questionnaire – Revised 18 (Karlsson et al., 2000), Eating Disorder Examination Questionnaire 6.0 (Fairburn, 2008), knowledge questionnaire, Dieting Intentions Scale (Cruwys et al., 2013), Weight Control Beliefs Questionnaire (Laliberte et al., 2007), Rosenberg Self-Esteem Scale (Rosenberg, 1989), and the Body Appreciation Scale – 2 (Tylka & Wood-Barcalow, 2015). Once the preliminary questionnaires are complete, the student investigator will project two educational videos. After watching the videos, participants will complete the following questionnaires on REDCap: knowledge questionnaire, Dieting Intentions Scale (Cruwys et al., 2013), Weight Control Beliefs Questionnaire (Laliberte et al., 2007), Rosenberg Self-Esteem Scale (Rosenberg, 1989), and Body Appreciation Scale – 2 (Tylka & Wood-Barcalow, 2015). At the end of the session, after watching the educational videos and completing the study questionnaires, participants will

receive a virtual copy of the debriefing form, which provides further information about the study purpose, independent and dependent variables, local mental health resources, and contact information for the LPI. The student investigator will review the debriefing form with the participants and provide an opportunity to ask any questions.

As stated above, if a participant does not present to the study appointment with an electronic device, the study team will provide the participant with a spare tablet to access and complete the study questionnaires on REDCap. As the questionnaires are completed on REDCap, no personal data will be stored on the tablet.

#### **Content and Development of Video Modules**

Each of the video modules provides evidence-based information on a particular topic: 1) weight science; 2) healthy nutrition; and 3) sleep hygiene. The weight science video discusses the research on the genetic contribution to body weight; the role of genetics in how individuals' body weight responds to over-eating; the research comparing the efficacy of different dieting approaches; the research on the long-term efficacy of behavioural approaches to weight loss; weight loss in obesity; research on the weight-loss registry looking at successful weight losers; and research on weight control beliefs. The healthy nutrition video discusses the development of food guides around the world; a definition and description of benefits of the "basics" of healthy eating (e.g., regular eating, balanced eating and pleasurable eating); a review of the macronutrients and their importance to health; a review of the recommendations concerning the specific food groups in the Canada's food guide; and how to put this all together to create a healthy eating plan. The sleep hygiene video, which is an active control, reviews the cognitive, emotional, physical health and weight implications of good quality sleep; provides a review of good sleep hygiene; and provides an overview of how to manage insomnia. The videos are all narrated by Dr. Michele Laliberte, a licensed clinical psychologist, and the information is consistent with current research and recommendations in the three areas discussed in the videos. There is no deception involved and it is made clear to participants that the information they are being provided is based on current research and the purpose is to understand the impact of this information on their attitudes and beliefs.

#### **Definition of end-point(s)**

The study will be published on SONA as soon as REB approval is granted. Data collection will continue until 150 participants are recruited. We anticipate collecting data from the start of January 2026 to August 2026. As McMaster University is offering first-level courses offerings in introductory psychology during this period, the investigators expect that it should be possible to recruit the targeted sample size within this timeframe.

#### Measurements and measurement instruments

The following self-report instruments will be used in the study:

- 1. Demographic Questionnaire
- 2. Three-Factor Eating Questionnaire Revised 18 (Karlsson et al., 2000)
- 3. Eating Disorder Examination Questionnaire 6.0 (Fairburn, 2008)
- 4. Knowledge Questionnaire
- 5. Dieting Intentions Scale (Cruwys et al., 2013)
- 6. Weight Control Beliefs Questionnaire (Laliberte et al., 2007)
- 7. Rosenberg Self-Esteem Scale (Rosenberg, 1989)
- 8. Body Appreciation Scale 2 (Tylka & Wood-Barcalow, 2015)

Study Link:

The online consent form and questionnaires may be accessed using the following link: <a href="https://edcredcap.mcmaster.ca/surveys/?s=YJ9HXWD97L7NDHPE">https://edcredcap.mcmaster.ca/surveys/?s=YJ9HXWD97L7NDHPE</a>

#### Data analysis plan

All analyses will be conducted in SPSS (version 27). In order to characterize the sample, descriptive statistics will be used. A multivariate analysis of variance (MANOVA) will be used to compare the three groups on change in weight control beliefs and eating pathology. Regression analyses will be used to look at the relationship between change in weight control beliefs and measures of eating pathology (dietary restraint, self-esteem, body appreciation, and the intent to diet) over the intervention. The regression analyses will be done across the entire sample.

#### How subjects will be recruited, including advertisements/publicity

All participants will be recruited through the McMaster University undergraduate psychology subject pool via SONA. The study will be advertised on the SONA on the "Study Sign-Up" page. A copy of the study advertisement can be found in Appendix A. On this page, potential participants are able to view the study title, a brief description of the study, compensation structure of the study, and study eligibility criteria. If a participant is interested in further information about the study, they are able to click on the study to learn the following about the study:

- 1. Study Name
- 2. Study Type
- 3. Credits (allocated for study completion)
- 4. Study Duration
- 5. Sign-Up Restrictions

- 6. Abstract
- 7. Study Description
- 8. Preparation
- 9. Eligibility Requirements
- 10. Website
- 11. Researcher Names & Contact Information
- 12. MREB Approval Code (HiREB Approval Code)

After considering all of the information relevant to the study, participants are able to sign-up for the study. This protocol allows participants to self-select for studies that they are interested in participating in, and limits potential undue pressure to participate from researchers, colleagues, supervisors, and others.

#### References

- Ackard, D. M., Fulkerson, J. A., & Neumark-Sztainer, D. (2007). Prevalence and utility of DSM-IV eating disorder diagnostic criteria among youth. *The International Journal of Eating Disorders*, 40(5), 409–417. https://doi.org/10.1002/eat.20389
- Barakat, S., McLean, S. A., Bryant, E., Le, A., Marks, P., National Eating Disorder Research Consortium, Touyz, S., & Maguire, S. (2023). Risk factors for eating disorders: findings from a rapid review. *Journal of eating disorders*, 11(1), 8. https://doi.org/10.1186/s40337-022-00717-4
- Cash, T. F., Phillips, K. A., Santos, M. T., & Hrabosky, J. I. (2004). Measuring "negative body image": Validation of the Body Image Disturbance Questionnaire in a nonclinical population. *Body Image*, 1(4), 363–372. https://doi.org/10.1016/j.bodyim.2004.10.001
- Cruwys, T., Platow, M. J., Rieger, E., & Byrne, D. G. (2013). The development and validation of the Dieting Intentions Scale (DIS). *Psychological assessment*, *25*(1), 264–278. https://doi.org/10.1037/a0030547
- Fairburn, C. G. (2008). Cognitive Behavior Therapy and Eating Disorders. Guilford Press.
- Jebeile, H., Gow, M. L., Baur, L. A., Garnett, S. P., Paxton, S. J., & Lister, N. B. (2019).

  Treatment of obesity, with a dietary component, and eating disorder risk in children and adolescents: A systematic review with meta-analysis. *Obesity Reviews*, 20(9), 1287-1298. https://doi.org/10.1111/obr.12866
- Kabakuş Aykut, M., & Bilici, S. (2022). The relationship between the risk of eating disorder and meal patterns in University students. *Eating and weight disorders : EWD*, *27*(2), 579–587. https://doi.org/10.1007/s40519-021-01179-4

- Karlsson, J., Persson, L., Sjöström, L., & Sullivan, M. (2000). Psychometric properties and factor structure of the Three-Factor Eating Questionnaire (TFEQ) in obese men and women. Results from the Swedish Obese Subjects (SOS) study. *International Journal of Obesity*, 24(12), 1715-1725. https://doi.org/10.1038/sj.ijo.0801442
- Laliberte, M. M., Balk, D., Tweed, S., Smith, J., & Ghai, A. (2014). The impact of education on weight control beliefs. *Ethnicity and Inequalities in Health and Social Care*, 7(2), 86–95. https://doi.org/10.1108/EIHSC-11-2013-0041
- Laliberte, M. M., & Lucibello, K. M. (2022). Weight control beliefs in the treatment of bingeeating disorder: Why might they matter? *International Journal of Eating Disorders*, 55(6), 820–825. https://doi.org/10.1002/eat.23713
- Laliberte, M. M., Newton, M., McCabe, R., & Mills, J. S. (2007). Controlling Your Weight

  Versus Controlling Your Lifestyle: How Beliefs about Weight Control Affect Risk for

  Disordered Eating, 10534\_2006\_9060\_Fig3\_HTML.gif Dissatisfaction and Self-esteem.

  Cognitive Therapy and Research, 31(6), 853–869. https://doi.org/10.1007/s10608-006-9104-z
- Mintz, L. B., & Betz, N. E. (1988). Prevalence and correlates of eating disordered behaviors among undergraduate women. *Journal of Counseling Psychology*, 35, 463–471. https://doi.org/10.1037/0022-0167.35.4.463
- Neumark-Sztainer, D. R., Wall, M. M., Haines, J. I., Story, M. T., Sherwood, N. E., & van den Berg, P. A. (2007). Shared risk and protective factors for overweight and disordered eating in adolescents. *American journal of preventive medicine*, *33*(5), 359–369. https://doi.org/10.1016/j.amepre.2007.07.031

- Patton, G. C., Selzer, R., Coffey, C., Carlin, J. B., & Wolfe, R. (1999). Onset of adolescent eating disorders: population based cohort study over 3 years. *BMJ (Clinical research ed.)*, 318(7186), 765–768. https://doi.org/10.1136/bmj.318.7186.765
- Piran, N., & Gadalla, T. (2007). Eating disorders and substance abuse in Canadian women: A national study. *Addiction (Abingdon, England)*, 102(1), 105–113. https://doi.org/10.1111/j.1360-0443.2006.01633.x
- Polivy, N., & Herman, C. P. (2002). Causes of eating disorders. *Annual Review of Psychology*, 53(1), 187–213.
  - https://www.annualreviews.org/doi/10.1146/annurev.psych.53.100901.135103
- Rosenberg, M. (1989). *Society and the Adolescent Self-Image* (Revised edition). Wesleyan University Press.
- Stice, E., Gau, J. M., Rohde, P., & Shaw, H. (2017). Risk factors that predict future onset of each DSM–5 eating disorder: Predictive specificity in high-risk adolescent females. *Journal of Abnormal Psychology*, 126(1), 38–51. https://doi.org/10.1037/abn0000219
- Stice, E., & Shaw, H. E. (2002). Role of body dissatisfaction in the onset and maintenance of eating pathology: A synthesis of research findings. *Journal of Psychosomatic Research*, 53(5), 985–993. https://doi.org/10.1016/s0022-3999(02)00488-9Tylka, T. L., & Wood-Barcalow, N. L. (2015). The Body Appreciation Scale-2: Item refinement and psychometric evaluation. *Body Image*, 12, 53–67. https://doi.org/10.1016/j.bodyim.2014.09.006
- Vartanian, L. R., & Herman, C. P. (2006). Beliefs about the determinants of body weight predict dieting and exercise behavior. *Eating Behaviors*, 7(2), 176-179. https://doi.org/10.1016/j.eatbeh.2005.08.009

# APPENDIX A: SONA ADVERTISEMENT FOR RECRUITMENT OF PARTICIPANTS

# Study #19334, McMaster SONA Advertisement, January 2026 PI: Dr. Keisha Gobin; Student Investigators: Mindy Tat, Sarah Potter

The information below will be displayed on the McMaster SONA platform. The HiREB approval information is listed under "Description" due to the format of the website.

| Study Type: Study Status: | Standard (lab) study. This is a standard lab study. To participate, sign up, and go to the specified location at the chosen time. Visible to participants: No |
|---|---|
| | Active study: No |
| Duration: | 120 minutes |
| Credits: | 2 |
| Abstract: | The Effects of Weight Science and Nutrition<br>Education on Weight Control Beliefs, Body<br>Image, Self-Esteem and Eating Patterns in<br>Undergraduate Dieters |
| Description: | If you consent to participate, you will attend an in-person study session in Room 403 at McMaster's Psychology Complex (PC-403). On the day of your appointment, please contact the lead student investigator, Mindy Tat, at tatm@mcmaster.ca and wait outside the PC-403 doors. During the session, you will be asked to watch two videos and answer a series of online questionnaires. The first set of questionnaires will ask you information about your gender, ethnicity, eating patterns, body image, weight control beliefs, intent to diet, self-esteem, and behaviours related to body image. After these questionnaires you will watch two educational videos related to living a healthy lifestyle. Finally, you will complete a second set of questionnaires about eating patterns, body image, weight control beliefs, intent to diet, self-esteem, and behaviours related to body image. |

| | T |
|---|---|
| | This study will ask questions about your eating patterns, body image, intent to diet, |
| | beliefs about weight, self-esteem, and |
| | behaviours related to body image. It is |
| | possible that you may experience mild |
| | discomfort when completing the |
| | questionnaires. You may skip any question |
| | you do not wish to answer or withdraw from |
| | the study at any time without penalty. |
| | The questionnaires and videos will take |
| | approximately 120 minutes to complete, and |
| | you will receive 2 credits for your |
| | participation in the study. All responses are |
| | private and confidential. |
| | This study has been reviewed by the |
| | Hamilton Integrated Research Ethics |
| | Board under Project #19334. |
| | Principal Investigator: Dr. Keisha Gobin |
| | Lead Student Investigator: Mindy Tat |
| | Student Co-Investigator: Sarah Potter |
| Eligibility Requirements: | To participate, you must be 18 years old or |
| Engionity Requirements. | older, restricting your eating to try and lose |
| | weight, self-identify as a woman, have normal |
| | (or corrected to normal) hearing and vision, |
| | and be a current undergraduate student at |
| | McMaster University. |
| Preparation: | You are asked to bring, if possible, your cell |
| | phone, laptop or tablet as the questionnaires |
| | can be completed online. If this is not |
| | possible, we will provide a spare electronic device for you to complete the consent form |
| | and questionnaires. |
| Participant Sign-Up Deadline: | 24 hours before the study is to occur |
| Researchers: | - |
| | Mindy Tat |